CLINICAL TRIAL: NCT01652300
Title: Oral Health Education in Pregnancy Promotes Knowledge,Attitude and Performance of Pregnant Women About Oral Health.
Brief Title: The Effect of Oral Health Education in Pregnancy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gonabad University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, NarjesBahriBinabaj, Instructor in midwifery education, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUMS
Record Dates: First submitted 2012-07-17; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Pregnancy
Keywords: Oral health; education; knowledge; attitude; performance
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test group (Experimental): For test group intervention was two educational sessions lasting 1 hour, focused on oral and dental health and especially on oral and dental health during pregnancy
  Interventions: Behavioral: two educational sessions
- control (Other): received no education
  Interventions: Behavioral: no education

INTERVENTIONS:
Behavioral: two educational sessions — The test group had two educational sessions lasting 1 hour, focused on oral and dental health and especially on oral and dental health during pregnancy
  Other Names: two educational sessions lasting 1 hour
  Arms: test group
Behavioral: no education — women in the control group received no education
  Other Names: women in the control group received no education
  Arms: control

SUMMARY:
Periodontal diseased during pregnancy are associated with many unpleasant prenatal consequences including preeclampsia, preterm labor, and low birth weight (LBW). Treatment of such diseases and observance of oral and dental hygiene may to some large extent prevent such consequences. Unfortunately previous studies have shown that pregnant women have very little knowledge of oral and dental health implications. Given the fact that pregnancy my be a unique opportunity to initiate correct hygienic behaviors in young women, this paper has focused on studying the effects of oral and dental health education during pregnancy.

In this single blind clinical trial study,140 pregnant women receiving care from Khaje Rabi Regional Health Center in Mashhad city who were members of a community based multi-center were chosen by systematic clustering methods and randomly allocated into test and control groups. After intervention, two questionnaires were completed for demographic and pregnancy details of the participants. Knowledge, health belief and health behavior were assessed before intervention. The test group had two educational sessions lasting 1 hour, focused on oral and dental health and especially on oral and dental health during pregnancy. women in the control group received no education. Knowledge, health belief and health behavior were assessed immediately after and one month after intervention of all participants. Analysis of data was done using SPSS, t-test and chi-square tests.

DETAILED DESCRIPTION:
In this clinical trial study,140 pregnant women receiving care from Khaje Rabi Regional Health Center in Mashhad city who were members of a community based multi-center were chosen by systematic clustering methods and randomly allocated into test and control groups. After intervention, two questionnaires were completed for demographic and pregnancy details of the participants. Knowledge, health belief and health behavior were assessed before intervention. The test group had two educational sessions lasting 1 hour, focused on oral and dental health and especially on oral and dental health during pregnancy. women in the control group received no education. Knowledge, health belief and health behavior were assessed immediately after and one month after intervention of all participants. Analysis of data was done using SPSS, t-test and chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Spoke Persian
* minimum education margin of primary school studies
* Gestational age between 12 and 32 weeks
* lacked any type of physical or mental problem
* lacked of any disease that could prevent from taking dental care

Exclusion Criteria:

* who did not attend the education sessions
* failed to complete the questionnaires
* receive any special education between post-test and stability test

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Score of KAP about oral health | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: narjes BahriBinabaj, Msc, Principal Investigator — GonabadMUM
Locations (1):
- Mums, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- See also: "Click here for more information about this study:"The Effect of Oral Health Education in Pregnancy" — http://www.mums.ac.ir